CLINICAL TRIAL: NCT07134478
Title: A Single-center, Open-label, Two-period, Fixed-sequence Clinical Study to Evaluate the Effect of Rifampicin on the Pharmacokinetics of HSK31858 in Healthy Subjects
Brief Title: Clinical Study to Evaluate the Effect of Rifampicin on the Pharmacokinetics of HSK31858 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK31858-105
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination drug; (Experimental): HSK31858 Tablets and Rifampicin Capsules
  Interventions: Drug: HSK31858 Tablets On the morning of Day 1, a single dose of HSK31858 tablets 40 mg will be administered. Rifampicin capsules After a 5-day washout period, a single dose of rifampicin capsules 600 mg wi

INTERVENTIONS:
Drug: HSK31858 Tablets On the morning of Day 1, a single dose of HSK31858 tablets 40 mg will be administered. Rifampicin capsules After a 5-day washout period, a single dose of rifampicin capsules 600 mg wi — HSK31858 Tablets On the morning of Day 1, a single dose of HSK31858 tablets 40 mg will be administered.
  Rifampicin capsules After a 5-day washout period, a single dose of rifampicin capsules 600 mg will be administered every morning from Day 6 to Day 14. On the morning of Day 15, rifampicin capsules 600 mg and HSK31858 tablets 40 mg will be co-administered.

SUMMARY:
This is a single-center, open-label, two-period, fixed-sequence clinical study to evaluate the effect of Rifampicin on the pharmacokinetics of HSK31858 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, aged 18 to 45 years (inclusive) at screening;
* Body weight ≥ 50 kg for males and ≥ 45 kg for females at screening; body mass index (BMI = weight (kg)/height2 (m2)) should be within the range of 19.0-26.0 kg/m2 (inclusive);
* Subjects (including their partners) agree to have no fertility plan, no sperm or egg donation plans, and take effective non-drug contraceptive measures (including complete abstinence, condoms, intrauterine device, partner sterilization, etc.) during the study and within 3 months after the last dose;
* Fully understand the purpose, requirements and potential risks of this study, voluntarily participate in the clinical study, and be able to sign the informed consent form (ICF) before the study;

Exclusion Criteria:

* Subjects with a known allergy to HSK31858 tablets, rifampicin capsules, or any component of similar drugs and preparations, or those with an allergic constitution (e.g., allergies to two or more drugs or food allergies); or those with a history of specific allergies (e.g., asthma, urticaria, eczema, etc.);
* Subjects who have special dietary requirements and cannot follow a uniform diet (including those with lactose intolerance); or those with dysphagia;
* Subjects with clinically significant abnormalities in vital signs, physical examination, laboratory tests (blood routine test, blood biochemistry, coagulation function, urinalysis), 12-lead ECG, chest X-ray (anteroposterior), or color ultrasonography, which are inappropriate for participation in this study as judged by the investigator;
* Subjects who have excessively consumed tea, coffee, or caffeinated beverages (more than 4 cups per day, 1 cup = 250 mL) within 3 months prior to screening; or who have consumed tea or any food or beverage containing caffeine (such as coffee, chocolate, etc.) within 48 hours prior to the first dose; or who do not agree to stop consuming tea, coffee or food or beverages containing caffeine during the study;
* Subjects who have consumed large amounts of grapefruit-rich beverages or food (such as grapefruit, grapefruit juice, grapefruit jam, etc.) within 14 days prior to screening; or who have consumed any grapefruit-rich beverages or food within 48 hours prior to the first dose; or who do not agree to stop consuming any grapefruit-rich beverages or food during the study;
* Subjects with a history or current diagnosis of significant cardiovascular, respiratory, digestive, urinary, hematological, endocrine, immune, dermatologic, or neurologic disease, including those who have undergone major surgery within 3 months prior to screening or whose surgical incision has not completely healed;
* Subjects with a history or current diagnosis of gastrointestinal, liver, kidney, or other diseases known to interfere with drug absorption, distribution, metabolism, or excretion;
* Subjects previously diagnosed with periodontitis or/and palmoplantar hyperkeratoses;
* Subjects who have donated or lost blood ≥ 400 mL within 3 months prior to screening or plan to donate blood during the study, or who have received blood transfusion or used blood products within 3 months prior to screening;
* Subjects who have used any drug that inhibits or induces hepatic CYP enzymes (e.g., CYP3A4 inducers-rifampicin, dexamethasone, carbamazepine, phenytoin, fosphenytoin, primidone, enzalutamide, St. John's Wort, etc.; CYP3A4 inhibitors-itraconazole, ketoconazole, voriconazole, erythromycin, clarithromycin, ritonavir, etc.) within 28 days prior to screening or within 5 half-lives of the drug (whichever is longer), or who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicine, or health care products other than those listed above within 14 days prior to screening or within 5 half-lives of the drug (whichever is longer);
* Subjects who have participated in other drug clinical studies within 3 months prior to screening; or who plan to participate in other clinical studies during the study;
* Subjects who have been vaccinated within 1 month before screening, or who plan to be vaccinated during the study;
* Subjects with a history of drug addiction, drug abuse, or drug dependence, or who have a positive drug abuse screening at screening;
* Subjects who have frequently consumed alcohol within 3 months before screening, that is, drinking more than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine), or who cannot abstain from alcohol during the study, or who have a positive breath alcohol test at screening;
* Subjects who have smoked more than 5 cigarettes per day (or equivalent amount of nicotine-containing products) within 3 months prior to screening, or who cannot abstain from smoking during the study;
* Subjects who are tested positive for one or more of the following at screening: hepatitis B virus surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, and Treponema pallidum antibody;
* Subjects with a history of needle sickness or blood sickness, difficulty in blood collection, or intolerance to blood collection by venipuncture;
* Subjects with tattoos or scars on any site of the skin that affect safety assessment as judged by the investigator;
* Women who are pregnant or breastfeeding; or those with a positive pregnancy test; Subjects who, in the investigator's opinion, have poor compliance or other factors that make them unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | [Time Frame: From the start of administration to 96 hours post-dose]
  The pharmacokinetic parameters of unchanged HSK31858 in plasma
AUC(0-∞) | [Time Frame: From the start of administration to 96 hours post-dose]
  The pharmacokinetic parameters of unchanged HSK31858 in plasma

SECONDARY OUTCOMES:
AUC(0-t) | [Time Frame: From the start of administration to 96 hours post-dose]
  The pharmacokinetic parameters of unchanged HSK31858 in plasma
Tmax | [Time Frame: From the start of administration to 96 hours post-dose]
  The pharmacokinetic parameters of unchanged HSK31858 in plasma
t1/2 | [Time Frame: From the start of administration to 96 hours post-dose]
  The pharmacokinetic parameters of unchanged HSK31858 in plasma
Cmax | [Time Frame: From the start of administration to 96 hours post-dose]
  The pharmacokinetic parameters of metabolite M4 in plasma
AUC(0-∞) | [Time Frame: From the start of administration to 96 hours post-dose]
  The pharmacokinetic parameters of metabolite M4 in plasma
Tmax | [Time Frame: From the start of administration to 96 hours post-dose]
  The pharmacokinetic parameters of metabolite M4 in plasma
AEs | [Time Frame: From the time of signing ICF to the end of follow-up，up to 25 days]
  The incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided